CLINICAL TRIAL: NCT05981196
Title: Individual and Structural-level Determinants Associated With Disparities Among Liver Transplant Patients
Brief Title: Disparities Among Liver Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adam J. Milam, Principal Investigator, Mayo Clinic
Other Study IDs: 22-008581
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-01

CONDITIONS: End Stage Liver DIsease
Keywords: Transplants; Transplantation; Healthcare Disparities; Minority Health; Communication
MeSH Terms: conditions — End Stage Liver Disease; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Liver Transplant Patients: Subjects with end-stage liver disease and being referred for transplant evaluation will fill out questionnaires about their background, emotions, and behaviors.

SUMMARY:
The purpose of this study is to inform healthcare interventions to reduce the disparities in liver transplant listing and in transplantation.

DETAILED DESCRIPTION:
Aim 1. Establish a longitudinal cohort of patients with end-stage liver dysfunction.

Aim 2. Examine interpersonal and structural factors associated with liver transplant evaluation and listing by patient characteristics (e.g., race, ethnicity, SES, gender).

Aim 3. Examine the use of stigmatizing language among patients undergoing liver transplant based on their demographic characteristics (e.g., race, ethnicity, SES, gender).

ELIGIBILITY:
Inclusion Criteria:

- Patients with end-stage liver, kidney, or cardiac dysfunction.

Exclusion Criteria:

* Patients with more than one system with end stage organ dysfunction, dementia, cognitive or sensory impairment, prior solid organ transplant.
* Patients with potential medical exclusions for transplant.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects identified with end-stage liver receiving initial stage of transplant evaluation at Mayo Clinic Arizona.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Liver transplant waiting list | Approximately one year
  Number of subjects listed on the liver transplant waiting list
Organ transplantation | Approximately one year
  Number of subject to receive an organ transplantation

SECONDARY OUTCOMES:
Survival | Approximately one year post-transplant, or until you are removed from the transplant list
  Total number of subject alive
Graft survival at six months | Six months post transplant
  Total number of subject to have a functioning graft at six months post transplant
Graft survival at one year | One year post transplant
  Total number of subject to have a functioning graft at one year post transplant

OTHER OUTCOMES:
Mortality | Approximately one year post-transplant, or until you are removed from the transplant list
  Total number of subject deaths
Hospital length of stay | Approximately one year post-transplant, or until you are removed from the transplant list
  Total number of days subjects were admitted to the hospital
ICU length of stay | Approximately one year post-transplant, or until you are removed from the transplant list
  Total number of days subjects were admitted to Intensive Care Unit (ICU)
30-day readmission | Approximately one year post-transplant, or until you are removed from the transplant list
  Number of subjects to experience a 30-day readmission

CONTACTS AND LOCATIONS:
Overall Officials: Adam Milam, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials